CLINICAL TRIAL: NCT05920668
Title: Phase IV Observational Study of Orelabrutinib in the Treatment of Chronic Lymphocytic Leukemia/Small Cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wang Xin (Other Government)
Responsible Party: Sponsor-Investigator, Wang Xin, Chief physician, Shandong Provincial Hospital
Organization: Shandong Provincial Hospital (Other Government)
Other Study IDs: CLL2023
Record Dates: First submitted 2023-06-05; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: CLL/SLL
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib monotherapy for CLL/SLL 12 cycles

SUMMARY:
This was a multicenter observational study of Orelabrutinib in the treatment of CLL/SLL. Patients were treated with Orelabrutinib for 12 cycles. The primary end points were grade 3 hypertension and incidence of atrial fibrillation, and the secondary end points were improvement in abnormal markers, ORR,CR,PFS, and OS.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-80 years old, gender unlimited; 2. Chronic lymphocytic/small cell leukemia was confirmed by histopathology based on iwCLL criteria; 3. According to the iwCLL standard, the treatment can be certified 4. IPI ≥ 2 5. ECOG score ≤2 points; 6. Measurable lesions detected by enhanced computed tomography/magnetic resonance imaging (CT/MRI) : at least one lymph node with a maximum axis of more than 1.5cm and a measurable vertical dimension; For patients with chronic lymphocytic leukemia, only peripheral circulating lymphocyte count must be required. 5000/μL (or 5×10^9/L); 7. If the major organs are functioning normally, the following criteria are met:

  1. The standard of blood routine examination shall meet:

     Neutrophil absolute value (ANC) ≥1.0×109/L, platelet (PLT) ≥30×109/L; Unless it is confirmed that the bone marrow and hematopoietic deficiency is caused by CLL/SLL;
  2. Biochemical examination shall meet the following standards:

TBIL < 2.0×ULN, CLL/SLL involved liver or diagnosed Gilbert syndrome (normal direct bilirubin), total bile red ≤ 3 ULN; ALT and AST < 2.5×ULN (for CLL/SLL involved liver, ALT and AST < 5×ULN); Endogenous creatinine clearance ≥30ml/min (Cockcroft-Gault formula). 8. Women of childbearing age must have been using reliable contraception or have had a pregnancy test (serum or urine) with negative results within 7 days prior to inclusion and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last test drug administration. For males, consent is required to use an appropriate method of contraception or surgical sterilization during the trial period and 8 weeks after the last administration of the trial drug; 9. Expected survival > 6 months; 10. Patients voluntarily participated in this study and signed written informed consent.

Exclusion Criteria:

* 1. Patients who have received other BTK inhibitors in the past and have progressed; 2. Patients with grade 3 hypertension 3. Patients with atrial fibrillation 4. Richter's syndrome is or has been confirmed by biopsy pathology; 5. Has active and uncontrolled autoimmune hemocytopenia, including autoimmune hemolytic anemia and idiopathic thrombocytopenic purpura; 6. Present or past malignancies other than cured basal cell carcinoma of the skin, carcinoma in situ of the cervix and superficial bladder carcinoma; 7. Received glucocorticoid therapy (at a dose of 20 mg/ day or higher than prednisone or equivalent) within 14 days prior to initial administration, except for inhalation, topical, intraarticular, and prophylactic use before or after use of iodized contrast agent; After discussion with the group leader, higher doses and longer steroid therapy may be permitted in the following situations:

  1. Treatment of autoimmune hemolysis or autoimmune thrombocytopenia associated with CLL/SLL disease;
  2. Short-term (within 14 days) use to treat non-active infections in diseases not associated with CLL/ SRL (e.g., arthritis, asthma) to acute exacerbations, including dose adjustments of steroids required for adrenal insufficiency; 8. Patients who have undergone major surgical operations (tests for diagnostic purposes) or participated in clinical trials of drugs/devices within 4 weeks; 9. Have uncontrolled or significant cardiovascular disease, including:

  <!-- -->

  1. New York Heart Association (NYHA) Class II or higher congestive heart failure, unstable angina, myocardial infarction, or arrhythmia requiring treatment at the time of screening, left ventricular ejection fraction (LVEF) &lt in the six months prior to the initial administration of the study drug; 50%;
  2. Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restricted cardiomyopathy, unestablished cardiomyopathy);
  3. Clinically significant history of prolonged QTc interphase, or women with interphase QTc in screening period > 470ms, male > 450ms;
  4. Subjects with symptomatic or medicated coronary heart disease;
  5. Patients with uncontrolled hypertension (on the basis of improving their life style, their blood pressure is still not up to the standard after more than 1 month with the application of reasonably tolerable enough 2 or more antihypertensive drugs (including diuretics), or their blood pressure can be effectively controlled by taking 4 or more antihypertensive drugs); 10. Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN+4 s or APTT > 1.5 ULN) or had active bleeding within 2 months prior to screening, or was taking anticoagulant drugs, or had what the investigator considered a definite tendency to bleed; 11. Arteriovenous thrombosis events, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc. occurred within 12 months before enrollment; 12. Clinically significant gastrointestinal abnormalities that may affect drug intake, transport, or absorption (e.g. inability to swallow, chronic diarrhea, intestinal obstruction, etc.); 13. Active or uncontrolled HBV (HBsAg positive and HBV DNA titer positive), HCV Ab positive or HIV positive; 14. Uncontrolled, active systemic fungal, bacterial, viral or other infection (defined as showing persistent signs/symptoms associated with the infection despite no improvement with appropriate antibiotics or other treatment); 15. Allergic disposition or hypersensitivity to obutinib or any other component of the applicable investigational drug; 16. Those who have received potent CYP3A4 inhibitor therapy within 7 days before enrollment, or potent CYP3A4 inducer therapy within 12 days before enrollment, or must also take CYP3A severely inhibiting or strongly inducible drugs; 17. Those who have a history of psychotropic substance abuse and cannot abstain or have mental disorders; 18. Participated in clinical trials of other antitumor drugs within 4 weeks before enrollment; 19. Pregnant and lactating women and subjects of childbearing age who do not want to take contraceptive measures; 20. Poor compliance or inability to follow up regularly; 21. Patients with life-threatening conditions or severe organ dysfunction are deemed unfit to participate in the study; 22. The investigator determines other circumstances that may affect the conduct of clinical studies and the determination of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:1. Age 18-80 years old, gender unlimited;2. Chronic lymphocytic/small cell leukemia was confirmed by histopathology based on iwCLL criteria;3. According to the iwCLL standard, the treatment can be certified 4.IPI ≥ 25. ECOG score ≤2 points; Exclusion Criteria:1. Patients who have received other BTK inhibitors in the past and have progressed;2. Patients with grade 3 hypertension 3. Patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of Grade 3 hypertension and atrial fibrillation | at the end of 12 cycles of treatment（(each cycle is 28 days)
  Number of patients with grade 3 or above hypertension during treatment/total number of patients enrolled; number of patients with atrial fibrillation during treatment/total number of patients enrolled.

SECONDARY OUTCOMES:
ORR | at the end of 12 cycles of treatment(each cycle is 28 days)
  Objective Response Rate
CR | at the end of 12 cycles of treatment(each cycle is 28 days)
  complete response
PFS | From the date of receipt of the first investigational medication to the date of first onset of disease progression or death from any cause, whichever comes first.up to 2 years
  progression-free survival
OS | From the date of receipt of the first study medication to the date of death from any cause.up to 2 years
  Overall Survival
Improvement rate of abnormal indicators | After 12 cycles of treatment(each cycle is 28 days)
  Continuous improvement in hematology (hemoglobin level increased to greater than 110g /L or ≥20 g/L increase from baseline, or platelet count increased to ≥50% from baseline, without blood transfusion/growth factors)
QoL | at the end of 12 cycles of treatment(each cycle is 28 days)
  Quality of Life score

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided